CLINICAL TRIAL: NCT01586052
Title: A Phase 1 Clinical Research of Erythropoietin Therapy for Children With Cerebral Palsy: Safety and Efficacy
Brief Title: Erythropoietin Therapy for Children With Cerebral Palsy: Phase 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPEPOPhase1
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Erythropoietin; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythropoietin and Rehabilitation (Experimental): recombinant human erythropoietin injection and active rehabilitation
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — 250 IU/kg, Twice a week for 4 weeks
  Other Names: Espogen produced by LG Life Science

SUMMARY:
This purpose of this phase 1 study is to investigate the safety and efficacy of erythropoetin for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a disorder of movement and posture resulted from a nonprogressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability.

Many experimental animal studies have revealed that erythropoietin is useful to repair neurological injury in brain. The main mechanism of erythropoietin is supposed as follows; neuroprotection effect, angiogenesis, and anti-inflammation.

On the basis of many experimental studies, erythropoietin is suggested as a potential therapy for cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* Abnormal Muscle Tone
* GMFCS (Gross Motor Functional Classification System): II to IV
* Age: 6 months ~ 3 years
* Abnormal Brain MRI compatible to clinical features and non-progressive
* Willing to Comply with All Study Procedure

Exclusion Criteria:

* Known Genetic Disorder
* Baseline Erythropoietin level > 45 mU/mL
* Presence of Drug Hypersensitivity Related to the Study Remedy
* Previous Erythropoietin Treatment before 3 months
* Coagulopathy:

Family History, Unknown Cerebral Infarction, Thromboembolic Events History

* Intractable Seizure Disorder
* Poor Cooperation of Guardian including Inactive Attitude for Rehabilitation
* Uncontrolled Hypertension
* Liver Dysfunction
* Renal Dysfunction
* Absolute Neutrophil Count < 500/dL
* Intracerebral or Intraventricular Hemorrhage
* Malignancy

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 8 weeks
  Monitoring of all adverse events during 8 weeks, the study period We selected specially considered adverse events: encephalopathy, intracranial hemorrhage, seizure, hypertension, thromboembolic event, hypoxia, and acute kidney injury. Other adverse events will be recorded. The list was determined by the clinical experience and all adverse reactions reported by the pharmaceutical company.

SECONDARY OUTCOMES:
Changes in Quality of Movement | Baseline - 8 weeks
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones: alignment, coordination, dissociated movement, stability, and weight shift The interrater reliability of GMPM subscores and total scores was 0.758-0.886 (subject n=75, tester n=10).
Changes in Gross Motor Function | Baseline - 8 weeks
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of 6 sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping The measured interrater reliability of GMFM subscores and total scores was 0.974 - 0.997 (subject n=101, tester n=10) and intrarater reliability of GMFM subscores and total scores between one most experienced rater and another newly t rained rater was 0.994 - 1.000 (subject n=101, tester n=2).
Changes in Neurodevelopmental Outcomes | Baseline - 8 weeks
  K-BSID-II (Korean version of Bayley Scale of Infant Development-II) Motor and Mental scales The measured intrarater and interrater reliability of K-BSID-II motor and mental scales was 0.92 - 0.99 (subject n=55, tester n=10).
Changes in Motor Development | Baseline - 8 weeks
  AIMS (Alberta Infant Motor Scale) to assess motor development
Changes in Spasticity | Baseline - 8 weeks
  MAS (modified Ashworth Scale) measured at biceps, hip adductor, hamstring, heel cord

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea